CLINICAL TRIAL: NCT06384430
Title: Subacromial Impingement Syndrome: The Relationship Between Shoulder Functional Tests and Ultrasound Parameters
Brief Title: Subacromial Impingement Syndrome Functional Tests Correlation With Ultrasound Parameters
Status: Recruiting | Type: Observational
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Nihal KARAYER OZGUL, Principal Investigator, Muğla Sıtkı Koçman University
Other Study IDs: MuğlaSKU-NKO
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Subacromial Impingement Syndrome; Shoulder Tendinitis; Shoulder Bursitis; Shoulder Pain
MeSH Terms: conditions — Shoulder Impingement Syndrome; Shoulder Pain | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with subacromial impingement syndrome: Patients with subacromial impingement syndrome: Being between 18-70 years old Clinical evaluation positive for subacromial impingement syndrome (Neer's test, Hawkins Kennedy, supraspinatus palpation test)
  Interventions: Diagnostic Test: Shoulder functional tests and ultrasound

INTERVENTIONS:
Diagnostic Test: Shoulder functional tests and ultrasound — On the day of the study, demographic data will be collected from patients with a clinical diagnosis of impingement and who agree to participate in the study, then DASH and Constant Murley scores will be calculated and subacromial bursa thickness, supraspinatus tendon thickness, acromiohumeral distance, supraspinatus tendon thickness/acromiohumeral distance ratio will be calculated on ultrasound.

SUMMARY:
In this study, among the patients who applied to the Physical Medicine and Rehabilitation outpatient clinic of Muğla Training and Research Hospital and were diagnosed with subacromial impingement by anamnesis and clinical tests, inclusion criteria) and exclusion criteria will be included in the study. Demographic data of the patients will then be recorded. DASH (Disabilities of the Arm, Shoulder and Hand) and Constant Murley scores will be calculated. 4 years of musculoskeletal ultrasound experience will be recorded by a radiologist using ultrasound (Siemens® V8, LA2-14A probe) in modified Crass position (positioning with the palm of the examined side on the posterior iliac wing) by measuring subacromial bursa thickness, supraspinatus tendon thickness, acromiohumeral distance, supraspinatus tendon thickness/acromiohumeral distance ratio. Demographic data of the patients will then be recorded. DASH (Disabilities of the Arm, Shoulder and Hand) and Constant Murley scores will be calculated.

DETAILED DESCRIPTION:
Subacromial impingement syndrome is a common shoulder pain disorder. In this study, among the patients who applied to the Physical Medicine and Rehabilitation outpatient clinic of Muğla Training and Research Hospital and were diagnosed with subacromial impingement by anamnesis and clinical tests, inclusion criteria (being between 18-70 years of age, positivity for subacromial impingement syndrome in clinical evaluation (Neer's test, Hawkins Kennedy, supraspinatus palpation test)) and exclusion criteria (under 18 years of age, over 70 years of age, rheumatologic disease diagnosis, symptomatic shoulder osteoarthritis, shoulder instability; shoulder pain in active, passive cervical spine movements, previous shoulder surgery, those with adhesive capsulitis findings (>50% passive range of motion restriction in 2 planes or full-thickness rotator cuff tear detected on ultrasound), those who received physiotherapy or intra-articular injections in the last 3 months, those with type 2 diabetes or hypothyroidism) will be included in the study. Demographic data of the patients will then be recorded. DASH (Disabilities of the Arm, Shoulder and Hand) and Constant Murley scores will be calculated. 4 years of musculoskeletal ultrasound experience will be recorded by a radiologist using ultrasound (Siemens® V8, LA2-14A probe) in modified Crass position (positioning with the palm of the examined side on the posterior iliac wing) by measuring subacromial bursa thickness, supraspinatus tendon thickness, acromiohumeral distance, supraspinatus tendon thickness/acromiohumeral distance ratio. Demographic data of the patients will then be recorded. DASH (Disabilities of the Arm, Shoulder and Hand) and Constant Murley scores will be calculated.

ELIGIBILITY:
Inclusion Criteria:

1. Being between 18-70 years old
2. Clinical evaluation positive for subacromial impingement syndrome (Neer's test, Hawkins Kennedy, supraspinatus palpation test)

Exclusion Criteria:

1. Under 18, over 70 years of age
2. Those diagnosed with rheumatologic diseases
3. Those with symptomatic shoulder osteoarthritis
4. Those with shoulder instability
5. Shoulder pain in active, passive cervical spine movements
6. Previous shoulder surgery
7. Findings of adhesive capsulitis (>50% restriction of passive range of motion in 2 planes or detection of a full-thickness rotator cuff tear on ultrasound)
8. Physiotherapy or intra-articular injection in the last 3 months
9. Diagnosis of type 2 diabetes or hypothyroidism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Being between 18-70 years old and clinical evaluation positive for subacromial impingement syndrome.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
subacromial bursa thickness | 1 day
  subacromial bursa thickness measure
supraspinatus tendon thickness | 1 day
  supraspinatus tendon thickness measure
acromiohumeral distance | 1 day
  acromiohumeral distance measure

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Egitim Arastima, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided